CLINICAL TRIAL: NCT02787096
Title: Dynamic Knee Laxity Measurement Coupled to MRI in Cases of Suspected Partial Anterior Cruciate Ligament Tear
Acronym: LaxIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-685
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: dynamic knee laxity measurement; laxi-MRI; partial anterior cruciate ligament tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laxIRM (Experimental): Patients will have dynamic knee laxity measurement coupled to MRI for the diagnosis of ACL tear
  Interventions: Device: LaxIRM

INTERVENTIONS:
Device: LaxIRM — Dynamic knee laxity measurement coupled to MRI for the diagnosis of ACL tear

SUMMARY:
Anterior cruciate ligament (ACL) tear is frequent, but the diagnosis of partial tears is difficult. Standard MRI may be used but is of limited diagnostic value. The present study aimed to evaluate the diagnostic interest of dynamic knee laxity measurement coupled to MRI for the diagnosis of ACL tear.

ELIGIBILITY:
Inclusion Criteria:

* knee injury requiring MRI examination
* accepting to participate
* covered by a health care insurance system

Exclusion Criteria:

* MRI contraindication
* pregnancy
* patient included in another study potentially affecting the results
* protected patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Anterior tibial translation (ATT) measurement | 1 year after the baseline MRI-scan
  Time Frame : 1 year after the baseline MRI-scan a follow-up MRI is performed if the patient did not had surgery.
  ATT is calculated as the difference between the distance from the tangent to the condyle to the tangent to the posterior aspect of the tibial plateau in the stress position and in resting conditions. ATT is measured for the medial and the lateral compartment respectively and the final ATT is the average of medial and lateral ATT.

SECONDARY OUTCOMES:
Degree of laxity | 1 year after the baseline MRI-scan
  1 year after the baseline MRI-scan a follow-up MRI is performed if the patient did not had surgery.
  Laxity of the torn ligament is defined using a visual scale with the following grading : 0 : No laxity. Grade 1: moderate laxity. Grade 2: severe laxity.
Femorotibial rotation (FTR) value | 1 year after the baseline MRI-scan
  1 year after the baseline MRI-scan a follow-up MRI is performed if the patient did not had surgery.
  FTR= arc tan ((ATT lateral-ATT medial)/(slice thickness*number of sagittal slices))*180/π

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste PIALAT, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot Pavillon B Radiologie, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pialat, Jean-Baptiste and Ltaief-Boudrigua, A. and Peyron, C. and Arion, S. and Manera, L. and Barta, A. Imagerie du genou : variantes à connaître, pièges à éviter. 44e Congrès thématique de la Société d'Imagerie Musculo-Squelettique - Le Genou. 2017-06-23/2017-06-24
- [Result] Lavigne, Joris and Stacoffe, Nicolas and Heidelberg, Damien and Pialat, Jean-Baptiste. 50 cas cliniques en radiologie pédiatrique ostéoarticulaire. Journées Francophones de Radiologie Diagnostique et Interventionnelle (JFR 2018) - 2018-10-12/2018-10-15